CLINICAL TRIAL: NCT03382106
Title: Smoking Cessation and Functional CT Assessment of Pulmonary Arterial Dysfunction in Smoking Associated Emphysema
Brief Title: Smoking Cessation and Functional CT Assessment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eric A. Hoffman (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Eric A. Hoffman, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 201706713; R01HL130883 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Emphysema
MeSH Terms: conditions — Emphysema | interventions — Sildenafil Citrate; Pulse Wave Analysis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subject and study team are masked to which arm subject is assigned (study drug or placebo). Investigational pharmacy will not be masked. For the non-smoker groups, both subjects and the study team will know which group they are assigned to (study drug or no medication).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Smoking Cessation Group 1 (Experimental): 80 normal smokers will be recruited (defined by Pulmonary Function Tests, questionnaires and interviews), between the ages of 21 and 65 will be studied to assess inflammation and heterogeneity of Perfused Blood Volume prior to and following a 3 month smoking cessation program. In 40 of the 80 subjects during the smoking cessation program, we will provide three times per day Sildenafil 20 milligrams (MG) (Viagra) for the full 3 months of the smoking cessation period. We select a three-month cessation program to maximize the likelihood of compliance with cessation yet providing enough time for a resolution of lung injury to take place. Pulse wave velocity, carotid artery compliance and stiffness and pressure wave reflection will be measured.
  Interventions: Drug: Sildenafil 20 MG; Diagnostic Test: Pulse wave velocity; Diagnostic Test: Carotid artery compliance and stiffness; Diagnostic Test: Pressure wave reflection
- Smoking Cessation Group 2 (Placebo Comparator): 80 normal smokers will be recruited (defined by Pulmonary Function Tests, questionnaires and interviews), between the ages of 21 and 65 will be studied to assess inflammation and heterogeneity of Perfused Blood Volume prior to and following a 3 month smoking cessation program. In 40 of the 80 subjects during the smoking cessation program, we will provide three times per day placebo oral tablet for the full 3 months of the smoking cessation period. We select a three-month cessation program to maximize the likelihood of compliance with cessation yet providing enough time for a resolution of lung injury to take place. Pulse wave velocity, carotid artery compliance and stiffness and pressure wave reflection will be measured.
  Interventions: Drug: Placebo Oral Tablet; Diagnostic Test: Pulse wave velocity; Diagnostic Test: Carotid artery compliance and stiffness; Diagnostic Test: Pressure wave reflection
- Non-Smokers Group 1 (Experimental): 20 non-smokers will be recruited (defined by Pulmonary Function Tests, questionnaires and interviews) between the ages of 21 and 65 will be studied to compare the heterogeneity of Perfused Blood Volume with that of smokers for a 3 month period of time. We will provide 10 females and 10 males three times per day Sildenafil 20 milligrams (MG) (Viagra) for the full 3 months.
  Interventions: Drug: Sildenafil 20 MG; Diagnostic Test: Pulse wave velocity; Diagnostic Test: Carotid artery compliance and stiffness
- Non-Smokers Group 2 (No Intervention): 20 non-smokers will be recruited (defined by Pulmonary Function Tests, questionnaires and interviews) between the ages of 21 and 65 will be studied to compare the heterogeneity of Perfused Blood Volume with that of smokers for a 3 month period of time. 10 females and 10 males will not receive any medication for the full 3 months.

INTERVENTIONS:
Drug: Sildenafil 20 MG — Sildenafil, 20mg three times daily for 3 month period.
  Other Names: Experimental: Smoking Cessation Group 1; Experimental: Non-Smokers Group 1
  Arms: Non-Smokers Group 1; Smoking Cessation Group 1
Drug: Placebo Oral Tablet — Placebo manufactured to look like Sildenafil 20 MG
  Other Names: No Intervention: Smoking Cessation Group 2
  Arms: Smoking Cessation Group 2
Diagnostic Test: Pulse wave velocity — Vascular pulse measurement at the radial, brachial, femoral, and carotid arteries are taken using a tonometer probe.
  Arms: Non-Smokers Group 1; Smoking Cessation Group 1; Smoking Cessation Group 2
Diagnostic Test: Carotid artery compliance and stiffness — An echocardiogram is done by using a probe placed on the skin.
  Arms: Non-Smokers Group 1; Smoking Cessation Group 1; Smoking Cessation Group 2
Diagnostic Test: Pressure wave reflection — Carotid pulse measurement taken using a tonometer probe
  Arms: Smoking Cessation Group 1; Smoking Cessation Group 2

SUMMARY:
The investigators will study the effect of pulmonary arterial vasodilation to see if it eliminates indices of persistent lung injury in smokers that are susceptible to emphysema.

DETAILED DESCRIPTION:
The purpose of this research study is to find out if smoking cessation combined with sildenafil, an FDA approved drug for pulmonary hypertension, will decrease inflammation in the lung. Even if a smoker stops smoking, the harmful effects caused by previous smoking may recruit inflammatory cells to those affected areas, leading to lung injury. In about 30-40% of smokers, this inflammation combined with irregular blood flow in the lungs may lead to emphysema. The study goal is to measure and compare individual responses to smoking cessation, Sildenafil and placebo used three times per day, and imaging of the lungs using non-contrast and contrast CT scans to see if there is a possible decrease of inflammation and an increase of blood flow in the lungs. The study also intends to see if using Sildenafil three times per day, in addition to smoking cessation will restore blood flow to the possible injured areas of the lungs. Sildenafil is an FDA approved medication for pulmonary hypertension but will be used off-label to study the effects it may or may not have on the blood flow in possible injured areas of the lungs. Non-smokers will be enrolled to compare lung imaging and the effects of Sildenafil on their lungs with that of smokers undergoing a smoking cessation program with placebo or Sildenafil. Non-smokers will complete identical measurements as smokers, with Sildenafil used three times per day or no medication across a similar 90 day period of time. Vascular measurements of pulse wave velocity, carotid artery compliance/stiffness and pressure wave reflection will be done at baseline and 90 day visits.

ELIGIBILITY:
Inclusion Criteria (Smokers):

* Between the age of 21 to 65 at baseline
* Be willing to participate in a smoking cessation program
* Be willing to attend all clinic visits
* Must be currently smoking at least ½ pack/day at baseline (confirmed with cotinine level and CO Smokerlyzer)
* >5 pack-year history of smoking
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) 0: FEV1≥0.80 and FEV1/FVC>0.70 Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC)
* GOLD 1: FEV1≥0.80 and FEV1/FVC < 0.70
* GOLD 2: 0.50≤FEV1<0.80 and FEV1/FVC < 0.70
* Be willing to abstain from using any nicotine patches, e-cigarettes, or marijuana for the duration of the study.

Inclusion Criteria (Non-smokers):

* Between the age of 21 to 65 at baseline
* Be willing to attend all clinic visits
* Have never smoked (confirmed with cotinine level and CO smokerlyzer)
* GOLD 0: FEV1≥0.80 and FEV1/FVC>0.70

Exclusion Criteria (Smokers and Non-smokers):

* Women only: Cannot be pregnant or nursing at baseline or plan to become pregnant during the course of the study
* Body Mass Index (BMI) > 35
* Allergies to shell fish, seafood, eggs or iodine
* Heart disease, kidney disease or diabetes
* Diagnosis of asthma
* Any metal in or on the body (that cannot be removed) between the nose and the abdomen
* Any major organ system disease (by judgment of the study medical team)
* A glomerular filtration rate of 60 cc per minute or less.
* Nitroglycerin usage or nitrates and use of phosphodiesterase 5 (PDE5) inhibitors
* Prior history of hypersensitivity to sildenafil
* Currently prescribed a phosphodiesterase (PDE) inhibitors medication (ex: Viagra, Cialis, etc)
* Known Pulmonary Hypertension
* Has used e-cigarettes and marijuana <1 years
* Use of ACE Inhibitors, Calcium Channel Blockers, Angiotensin II Receptor Blockers for control of blood pressure or any combination of these three types of medications.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Measure and compare individual smokers' responses to smoking cessation, Sildenafil and placebo with lung imaging to determine decrease of inflammation and increase of blood flow in lungs. | 90 Days
  Our outcome measure is the change in regional blood volume between baseline and interventions with CT imaging, sildenafil/placebo and smoking cessation.

SECONDARY OUTCOMES:
Pulse wave velocity of carotid radial, brachial, femoral and carotid arteries | Baseline and 90 day
  Our outcome measure is the difference of arterial stiffness between baseline and 90 day visits.
Carotid beta-stiffness index | Baseline and 90 Day
  Our outcome measure is the difference of common carotid artery stiffness between baseline and 90 day visits
Carotid augmentation index | Baseline and 90 Day
  Our outcome measure is the difference of pressure wave reflection between baseline and 90 day visits

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hoffman, PhD, Principal Investigator — Professor
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
CT images will be shared including non-contrast images at TLC, FRC and RV as well as dual energy CT image data used to assess regional perfused blood volume. All associated pulmonary function test results will be shared. CT-derived metrics.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available starting 6 months after publication of the primary results of each aim.
Access Criteria: Data will be provided to academic-based researchers upon written request to the PI, Eric A. Hoffman, PhD. A nominal charge will be made for the time it takes for a technician to prepare and transfer the requested data. These costs will not exceed $250. This service will be available for a minimum of 2 years of study close.

DOCUMENTS (2):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03382106/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT03382106/SAP_002.pdf